CLINICAL TRIAL: NCT04678570
Title: The Effect of White Noise and Swaddling Methods in Reducing the Pain Caused by Orogastric Tube Insertion in Preterm Infants: A Randomized Controlled Trial
Brief Title: Pain Perception Associated With Orogastric Tube Insertion in Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, ÖZNUR GÜRLEK KISACIK, Assistant Professor PhD, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-467
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-01

CONDITIONS: Orogastric Tube Insertion
Keywords: Pain; Preterm birth
MeSH Terms: conditions — Pain; Premature Birth

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The same nurse, who will perform the insertion of the orogastric tube, will be blinded to the control and the intervention groups.
  Another nurse, who will take the measurements of the heart rate and the saturation, will be blinded to the control and the intervention groups.
  2 observers, independent from the study, who will assess the pain will be blinded to the intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Group-1 (Experimental): White Noise intervention and standard care, procedures will be applied.
  Interventions: Other: White Noise
- Intervention Group- 2 (Experimental): The swaddling method and standard care, procedures will be applied.
  Interventions: Other: Swaddling Method
- Intervention Group- 3 (Experimental): White Noise, swaddling method, and standard care, procedures will be applied.
  Interventions: Other: White Noise; Other: Swaddling Method
- No Intervention Group (No Intervention): Standard care and procedures to be applied.

INTERVENTIONS:
Other: White Noise — The infants will be listened to a song Called " Bebeginiz Aglamasin" from Orhan Osman's colic album which was prepared with the help of Dr. Harvery Karp's ''The Happiest Baby'' album through a portable speaker located at 50 cm away from the infant at 55-decibel frequency.
  Listening to this song will start 5 minutes before the insertion of the Orogastric Tube, will continue during the procedure and another 5 more minutes after the procedure is completed. The rest of the noise in the environment will be controlled.
  Arms: Intervention Group- 3; Intervention Group-1
Other: Swaddling Method — The preterm infants will be placed in the supine position on a 90 cm2 soft cloth. The upper edge of the cloth will be aligned with the infant's shoulder, with the arms placed close to the body, with the horizontal ends of the cloth folded in the opposite direction to cover the top of the body. The arms will be put into flexion and the body will be covered with a cloth. In order not to limit the movements of all limbs of the preterm infant, attention will be paid to leave a finger space between the infant and the cloth cover and to leave a suitable space for the feet to be comfortable before folding the lower part of the cloth cover forward. In the swaddling method, the baby's head can move freely. The swaddling method will be applied approximately 5-10 minutes before the procedure and will be removed from the infant 5 minutes after the procedure. Because swaddling will increase the body temperature of the infant, the standard temperature of the incubator will be lowered.
  Arms: Intervention Group- 2; Intervention Group- 3

SUMMARY:
This study is a randomized controlled experimental study designed to examine the effect of white noise and swaddling methods in reducing the pain caused by orogastric tube insertion in preterm infants.

This study is planned to be conducted with 4 groups, consisting of 3 experimental groups and 1 control group. White noise, swaddling method, and white noise + swaddling methods will be the interventions during the study together with the standard care and procedures for the experimental groups, while the control group will only have standard care and procedures during the study.

DETAILED DESCRIPTION:
This is a randomized controlled experimental study designed to examine the effect of white noise and swaddling methods in reducing the pain caused by orogastric tube insertion in preterm infants.

The study will be conducted between 01/01/2021-15/06/2021 in Usak Öztan Hospital Neonatal Intensive Care Unit.

The sample of the study is planned to have 132 participants with 33 of them in each of the 4 groups.

This study is planned to be conducted with 4 groups, consisting of 3 experimental groups and 1 control group. White noise, swaddling method, and white noise + swaddling methods will be the interventions during the study together with the standard care and procedures for the experimental groups, while the control group will only have standard care and procedures during the study.

The interventions that will be used in this study are emphasized in the literature as nonpharmacological methods in reducing and preventing pain.

In Usak Öztan Hospital Neonatal Intensive Care Unit, where the study is planned to be conducted, a pre-application will be performed with 10 preterm infants to evaluate the effect of white noise, swaddling, white noise, and swaddling methods on pain perception in preterm infants with an orogastric tube inserted.

As the video recordings will be used for the evaluation of the pain, the best area for the video recorder to be placed will be decided during this stage.

Insertion of the orogastric tube will be done by the same nurse, who will be briefed about the study concept and will be blinded to the control and the intervention groups, to manage standardization. There will be always a specialist doctor to monitor the infants during this stage for any possible complications.

ELIGIBILITY:
Inclusion Criteria:

* With 32-34 weeks of gestation,
* With the postnatal age between 3-28 days,
* Birth weight is above 1000 grams,
* With the Apgar score ≥7 at 1st and 5th minutes,
* With stable vital signs,
* Without any congenital anomaly,
* Not receiving mechanical ventilator support and having spontaneous breathing,
* Requested by the physician to place an orogastric tube and fed with an orogastric tube,
* Breastfeeding (through an orogastric tube),
* Not experienced a painful procedure at least half an hour before the interventions,
* Without the use of opioid or non-opioid analgesic in their treatment,
* Without congenital or acquired malformation related to hearing,
* With parents written consent for the participation of their baby.

Exclusion Criteria:

* With the postnatal age outside 3-28 days,
* Birth weight is ≤ 1000 grams,
* With the Apgar score <7 at 1st and 5th minutes,
* With unstable vital signs,
* With congenital anomaly in the face or the oral cavity,
* Being on mechanical ventilator support,
* With a congenital malformation that may affect respiration and cause asphyxia,
* With intracranial bleeding or risk of bleeding,
* With disorders affecting the cerebral circulation or cardiovascular system,
* Subjected to a painful procedure at least half an hour before the interventions,
* With opioid or non-opioid analgesic in their treatment,
* With the surgical history,
* With continuous sedative treatment,
* With congenital or acquired malformation related to hearing,
* Not being fed with an orogastric tube,
* With parent not giving consent for the participation of their baby

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
The Premature Infant Pain Profile-Revised (PIPP-R) Change | 5 minutes, 3 minutes and 1 minute before the procedure. During the procedure. 1 minute, 3 minutes and 5 minutes after the procedure
  The PIPP-R scale includes 3 behavioral (brow bulge, eye squeeze, nasolabial-furrow), 2 physiological (heart rate and oxygen saturation) and 2 contextual (behavioral state and gestational age) items. Each item has a score from 0-3. The highest score that can be obtained from the PIPP-R scale for preterm infants is 21.The mean scores obtained from the PIPP-R scale reflects mild level of pain as mild if it is between 0-6 points, moderate if it is between 7-12 points and severe if it is between 13-21 points.

CONTACTS AND LOCATIONS:
Overall Officials: Öznur GÜRLEK KISACIK, Phd, Study Director — Afyonkarahisar Health Sciences University
Locations (1):
- Uşak Öztan Hospital Neonatal Intensive Care Unit, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No